CLINICAL TRIAL: NCT06322719
Title: A Randomized Comparison Between the Hyperangulated vs. Macintosh Blades for First-attempt Intubation Success With Videolaryngoscopy in ICU Patients.
Brief Title: Hyperangulated vs Macintosh Blades for Intubation With Videolaryngoscopy in ICU
Acronym: INVIBLADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Professor Anesthesiology, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INVIBLADE
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure; Intubation; Intubation; Difficult or Failed; Videolaryngoscopy; Intubation Complication
Keywords: videolaryngoscopy; tracheal intubation; complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperangulated videolaryngoscope (Experimental): Tracheal intubation facilitated by a hyperangulated videolaryngoscope
  Interventions: Device: Hyperangulated blade videolaryngoscope
- Macintosh videolaryngoscope (Active Comparator): Tracheal intubation facilitated by a videolaryngoscope with a Macintosh type blade
  Interventions: Device: Macintosh blade videolaryngoscope

INTERVENTIONS:
Device: Hyperangulated blade videolaryngoscope — For patients assigned to the Hyperangulated videolaryngoscope Group, the operator will use a Hyperangulated video laryngoscope on the first laryngoscopy attempt.
  Arms: Hyperangulated videolaryngoscope
Device: Macintosh blade videolaryngoscope — For patients assigned to the Macintosh videolaryngoscope Group, the operator will use a Hyperangulated video laryngoscope on the first laryngoscopy attempt.
  Arms: Macintosh videolaryngoscope

SUMMARY:
Tracheal intubation in the intensive care unit (ICU) is associated with high incidence of difficult intubation and complications. Videolaryngoscopes (VLs) devices have been proposed to improve airway management, and the use of VLs are recommended as first-line or after a first-attempt failure using direct laryngoscopy in ICU airway management algorithms. Although until relatively few years ago there were doubts about whether videolaryngoscopes had advantages over direct laryngoscopy for endotracheal intubation (ETI) in critically ill patients, two recent studies (DEVICE (1), INTUBATE (2)), and a Cochrane review (3) have confirmed that videolaryn should be used?, and what is the best blade? . There are two types of blades commonly used with videolaryngoscopes: the "Macintosh" blade with a slight curvature, and hyperangulated blades. The "Macintosh" blades have a lower angle of vision, but they have the advantage of being similar to the blades commonly used in direct laryngoscopy, making them easy to use for the person performing the ETI. Hyperangulated blades have a greater angle of vision, improving glottic visualization, especially in patients with an anterior glottis. However, the need to overcome this angulation could potentially hinder the passage of the endotracheal tube to the vocal cords. It is unknown if either blade has any advantage for intubating critically ill patients.

DETAILED DESCRIPTION:
The purpose of this prospective multicenter randomized study is to compare successful intubation on the first attempt with the Macintosh videolaryngoscope vs the hyperangulated videolaryngoscope during tracheal intubation in ICU patients.The hypothesis of the study is that tracheal intubation using the hyperangulated videolaryngoscope will improve the frequency of successful intubation on the first attempt in ICU patients requiring intubation in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Admitted to an Intensive Care Unit.
* Need for tracheal intubation during the stay in the ICU.
* The device to be used for intubation is a videolaryngoscope

Exclusion Criteria:

* Pregnancy or lactation.
* Emergent tracheal intubation that does not allow for the randomization of the procedure.
* Need for tracheal intubation with a device other than the videolaryngoscope (fiberoptic bronchoscope, direct laryngoscopy, tracheostomy, etc.).
* Tracheal intubation performed outside the ICU (Emergency Department, Hospital ward, etc.).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the first attempt intubation success rate (percentage) | During intubation (minutes)
  The primary outcome is defined as placement of an endotracheal tube in the trachea with a single insertion of a videolaryngoscope blade into the mouth and either a single insertion of an endotracheal tube into the mouth or a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube over the bougie into the mouth.

SECONDARY OUTCOMES:
Difference in the overall success rate | During intubation (minutes)
  To compare the difference overall success rate (percentage) with the two (hyperangulated vs Macintosh blades) videolaryngoscopes
Number of intubation attempts | During intubation (minutes)
  To compare number of intubations attempts with the two (hyperangulated vs Macintosh blades) videolaryngoscopes
Modified Cormack-Lehane grade of glottic view | During intubation (minutes)
  To compare Cormack-Lehane grade of glottic view with the two (hyperangulated vs Macintosh blades) videolaryngoscopes.
  Modified Cormack-Lehane grade of glottic view is defined as:
  Grade I: full view of the glottis Grade IIa: partial view of the glottis Grade IIb: arytenoid or posterior part of the vocal cords just visible Grade III: only epiglottis visible Grade IV: neither glottis nor epiglottis visible Cormack-Lehane grade of glottic view
Diference in the incidence of "easy intubation" | During intubation (minutes)
  To compare the difference in the incidence of "easy intubation" defined as a patient with Cormack-Lehane I-II glottic view and intubation on the first attempt.
Duration of tracheal intubation | Duration of procedure (minutes)
  To compare the interval (in seconds) between the first insertion of a videolaryngoscope blade into the mouth and the final placement of an endotracheal tube in the trachea.
Reason for unsuccessful intubation on the first attempt | Duration of procedure (minutes)
  Causes of unsuccessful intubation on the first attempt:
  * Limited visibility of the larynx
  * Difficulty in properly inserting the endotracheal tube
  * Challenges in cannulating the trachea with a bougie
  * Interruption of the attempt due to changes in the patient's condition (such as deteriorating hypoxemia, hypotension, bradycardia, vomiting, or bleeding)
  * Technical malfunctions with the laryngoscope equipment (such as battery issues, light source malfunction, camera problems, or screen issues)
  * Other factors
Number of videolaryngoscopy attempts | Duration of procedure (minutes)
  To compare the number of videolaryngoscope attempts neccesary to successfull tracheal intubation
Number of attempts to cannulate the trachea with a bougie or an endotracheal tube | Duration of procedure (minutes)
  To compare the number of attempts to cannulate the trachea with a bougie or an endotracheal tube
Operator-assessed difficulty of intubation | Duration of procedure (minutes)
  To compare operator-assessed subjective difficulty of intubation:
  * without difficulty
  * mild difficulty
  * moderate difficulty
  * severe difficulty
Need for additional airway equipment | Duration of procedure (minutes)
  Airway equipment: bougie, stylet, other videolaryngoscope, others
Need to change the device for intubation | Duration of procedure (minutes)
  Need to replace by another videolaryngoscope, a different angled blade, requirement for a fiberoptic bronchoscope...).
Complications of tracheal intubation | Duration of procedure (minutes)
  Complications:
  * Hypoxemia (lowest oxygen saturation measured by pulse oximetry 80%-90%)
  * Severe hypoxemia (lowest oxygen saturation measured by pulse oximetry < 80%)
  * Hypotension (systolic blood pressure between 80-65 mm Hg)
  * Severe hypotension (systolic blood pressure < 65 mm Hg)
  * Pulmonary aspiration
  * Esophageal intubation
  * Dental injuries
  * Airway injuries
  * Others

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada, Ph.D., Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (29):
- Spain (29):
  - University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña
  - Complexo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital General de Albacete, Albacete
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario de Cáceres, Cáceres
  - Hospital de Denia, Denia
  - Hospital General Universitario de Eche, Elche
  - Hospital Universitario de Cabueñes, Gijón, Gijón
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Majadahonda
  - Hospital Universitario de Móstoles, Móstoles
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Oviedo
  - Clínica Universidad de Navarra, Pamplona, Pamplona
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Donostia, San Sebastián, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander, Santander
  - Complejo Asistencial de Segovia, Segovia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
  - Complexo Hospitalario Universitario Álvaro Cunqueiro de Vigo, Vigo
  - Hospital Ribera Povisa Vigo, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Taboada M, Doldan P, Calvo A, Almeida X, Ferreiroa E, Baluja A, Carinena A, Otero P, Caruezo V, Naveira A, Otero P, Alvarez J. Comparison of Tracheal Intubation Conditions in Operating Room and Intensive Care Unit: A Prospective, Observational Study. Anesthesiology. 2018 Aug;129(2):321-328. doi: 10.1097/ALN.0000000000002269. PMID 29787386
- [Background] Higgs A, McGrath BA, Goddard C, Rangasami J, Suntharalingam G, Gale R, Cook TM; Difficult Airway Society; Intensive Care Society; Faculty of Intensive Care Medicine; Royal College of Anaesthetists. Guidelines for the management of tracheal intubation in critically ill adults. Br J Anaesth. 2018 Feb;120(2):323-352. doi: 10.1016/j.bja.2017.10.021. Epub 2017 Nov 26. PMID 29406182
- [Background] Prekker ME, Driver BE, Trent SA, Resnick-Ault D, Seitz KP, Russell DW, Gaillard JP, Latimer AJ, Ghamande SA, Gibbs KW, Vonderhaar DJ, Whitson MR, Barnes CR, Walco JP, Douglas IS, Krishnamoorthy V, Dagan A, Bastman JJ, Lloyd BD, Gandotra S, Goranson JK, Mitchell SH, White HD, Palakshappa JA, Espinera A, Page DB, Joffe A, Hansen SJ, Hughes CG, George T, Herbert JT, Shapiro NI, Schauer SG, Long BJ, Imhoff B, Wang L, Rhoads JP, Womack KN, Janz DR, Self WH, Rice TW, Ginde AA, Casey JD, Semler MW; DEVICE Investigators and the Pragmatic Critical Care Research Group. Video versus Direct Laryngoscopy for Tracheal Intubation of Critically Ill Adults. N Engl J Med. 2023 Aug 3;389(5):418-429. doi: 10.1056/NEJMoa2301601. Epub 2023 Jun 16. PMID 37326325
- [Background] Russotto V, Myatra SN, Laffey JG, Tassistro E, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Pelosi P, Sorbello M, Higgs A, Greif R, Putensen C, Agvald-Ohman C, Chalkias A, Bokums K, Brewster D, Rossi E, Fumagalli R, Pesenti A, Foti G, Bellani G; INTUBE Study Investigators. Intubation Practices and Adverse Peri-intubation Events in Critically Ill Patients From 29 Countries. JAMA. 2021 Mar 23;325(12):1164-1172. doi: 10.1001/jama.2021.1727. PMID 33755076
- [Background] Russotto V, Lascarrou JB, Tassistro E, Parotto M, Antolini L, Bauer P, Szuldrzynski K, Camporota L, Putensen C, Pelosi P, Sorbello M, Higgs A, Greif R, Grasselli G, Valsecchi MG, Fumagalli R, Foti G, Caironi P, Bellani G, Laffey JG, Myatra SN; INTUBE Study Investigators. Efficacy and adverse events profile of videolaryngoscopy in critically ill patients: subanalysis of the INTUBE study. Br J Anaesth. 2023 Sep;131(3):607-616. doi: 10.1016/j.bja.2023.04.022. Epub 2023 May 17. PMID 37208282
- [Background] Hansel J, Rogers AM, Lewis SR, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adults undergoing tracheal intubation: a Cochrane systematic review and meta-analysis update. Br J Anaesth. 2022 Oct;129(4):612-623. doi: 10.1016/j.bja.2022.05.027. Epub 2022 Jul 9. PMID 35820934
- [Background] Araujo B, Rivera A, Martins S, Abreu R, Cassa P, Silva M, Gallo de Moraes A. Video versus direct laryngoscopy in critically ill patients: an updated systematic review and meta-analysis of randomized controlled trials. Crit Care. 2024 Jan 2;28(1):1. doi: 10.1186/s13054-023-04727-9. PMID 38167459
- [Derived] Taboada M, Estany-Gestal A, Fernandez J, Vazquez O, Pajares A, Ramasco F, Martinez S, Vallejo I, Perez A, Rama-Maceiras P, Bermudez M, Power M, Garcia-Alvarez R, Fernandez-Villa I, Aguilera JL, Carrio M, Cabadas R, Rubin A, Williams MM, Fernandez-Garcia R, Becerra A, Gine M, Garcia FJ, Iglesias MC, Santamarina RM, Del Valle S, Charco LM, Alonso MC, Rodriguez IM, Varela M, Hermoso JI, Vives M, Cabaleiro T. Hyperangulated versus Macintosh blades for intubation with videolaryngoscopy in ICU: the randomised multicentre INVIBLADE-ICU trial study protocol. BMJ Open. 2024 Sep 5;14(9):e086691. doi: 10.1136/bmjopen-2024-086691. PMID 39237284